CLINICAL TRIAL: NCT04218422
Title: Battlefield Acupuncture to Treat Pain in Hidradenitis Suppurativa
Brief Title: Battlefield Acupuncture for Pain in Hidradenitis Suppurativa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Steven D Daveluy, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-19-12-1642
Record Dates: First submitted 2019-12-27; First posted 2020-01-06 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Hidradenitis Suppurativa
Keywords: acupuncture; pain; battlefield acupuncture; hidradenitis
MeSH Terms: conditions — Hidradenitis Suppurativa; Pain; Hidradenitis

STUDY DESIGN:
Intervention Model Description: Blinded, randomized trial
Who Masked: Participant
Masking Description: Participants will not know whether they got battlefield acupuncture or sham acupuncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): 2 treatments of battlefield acupuncture to the bilateral ears spaced one week apart
  Interventions: Procedure: Battlefield Acupuncture
- Control (Sham Comparator): 2 treatments with sham acupuncture to the bilateral ears at acupuncture points not associated with pain relief (2 liver and 1 stomach)
  Interventions: Procedure: Sham Acupuncture

INTERVENTIONS:
Procedure: Battlefield Acupuncture — Acupuncture at 5 points on the ears
  Arms: Treatment
Procedure: Sham Acupuncture — Sham acupuncture in 2 points for liver and 1 point for stomach
  Arms: Control

SUMMARY:
The investigators will investigate battlefield acupuncture as a treatment for the pain of hidradenitis suppurativa.

DETAILED DESCRIPTION:
Participants will report their pain level daily for 4 weeks. At week 2 and 3, they will get acupuncture in the ears.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* dermatologist-confirmed diagnosis of hidradenitis suppurativa
* significant pain from hidradenitis at least twice weekly
* stable treatment regimen for hidradenitis during study period

Exclusion Criteria:

* disease or disfigurement of the ear that prevents battlefield acupuncture of the ears
* other chronic pain that will interfere with the ability to rate hidradenitis pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2030-12-23 (Estimated); Study Completion 2031-02-20 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Numerical Rating Score | Average Score from scores Recorded daily for 4 weeks
  Difference in Average Patient self-reported Pain Numerical Rating Score from 0-10, comparing average from 2 weeks prior to treatment with average from 2 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- WSUPG Dermatology, Dearborn, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data

REFERENCES:
- [Background] Horvath B, Janse IC, Sibbald GR. Pain management in patients with hidradenitis suppurativa. J Am Acad Dermatol. 2015 Nov;73(5 Suppl 1):S47-51. doi: 10.1016/j.jaad.2015.07.046. PMID 26470616